CLINICAL TRIAL: NCT07161193
Title: Anti-CD19 Chimeric Antigen Receptor T Cells for Refractory Autoimmune Diseases
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, China (Unknown); Henan Province Engineering Technology Research Center of Immunological Precision Medicine and Artificial Intelligence Application, Luoyang, China (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L2025021-2
Record Dates: First submitted 2025-08-19; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Autoimmune Diseases
Keywords: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental :CD19 CAR (Experimental): Following the lymphodepleting treatment, patients will be treated with CD19 Chimeric Antigen Receptor (CAR) positive T cells as a single dose.
  Interventions: Biological: CD19 CAR-T cells

INTERVENTIONS:
Biological: CD19 CAR-T cells — Following lymphodepletion with chemotherapy (cyclophosphamide and fludarabine) patients will be treated with CD19 Chimeric Antigen Receptor (CAR) positive T cells as a single dose.

SUMMARY:
The goal of this study is to evaluate the safety and efficacy of CD19 CAR T cells in the treatment of Refractory Autoimmune Diseases

DETAILED DESCRIPTION:
This is a single-center, open-label, single-arm, dose-escalation trial. In this study, we will recruit seven kinds of refractory autoimmune diseases including moderate-to-severe Systemic lupus erythematosus (SLE), refractory Pemphigus, refractory Idiopathic inflammatory myopathy (IIM), Systemic sclerosis (SSc), Refractory ANCA-Associated Vasculitis/Nephritis,refractory Rheumatoid arthritis(RA) and moderate-to-severe refractory Psoriasis.

Patients with Refractory Autoimmune Diseases will receive CD19 CAR T cells. The primary objective is to evaluate the safety and efficacy of CD19 CAR T cell therapy in subjects with Refractory Autoimmune Diseases and to determine the optimal biological dose (OBD) in phase I and to learn about the efficacy CD19 CAR T-cell therapy in patients with Refractory Autoimmune Diseases in phase II.

The primary endpoint is to evaluate the incidence and severity of cytokine release syndrome and severe neurotoxic adverse events within 28 days after CAR-T cell infusion.A total number of 3o subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 1.Refractory Moderate-to-Severe Systemic lupus erythematosus (SLE) 1.1.Age 18-70 years. 1.2.Estimated life expectancy ≥ 3 months. 1.3.Documented disease history and diagnosis for ≥ 6 months prior to screening. 1.4.Participants must agree to use effective contraception throughout the study; women of child-bearing potential must have a negative pregnancy test.

1.5.Signed informed consent, agreement to the treatment protocol, and willingness to attend follow-up evaluations per schedule.

1.6.Relevant medical history and clinical manifestations: provide a copy of inpatient records from a tertiary hospital or outpatient records and diagnostic certificates within the last 3 months.

1.7.Required laboratory tests, including but not limited to: CBC, urinalysis, ANA, anti-dsDNA, ENA panel, C3/C4, immunoglobulins, antiphospholipid antibodies, etc.

1.8.Meets current international or domestic classification criteria: the 1997 ACR SLE classification criteria OR the 2019 EULAR/ACR SLE classification criteria, and is judged to have moderate-to-severe SLE.

1.9.SELENA-SLEDAI score ≥ 8; PGA ≥ 1; and at least one BILAG-2004 organ-system score of 1A or 2B.

1.10.Inadequate response to, or intolerance of, at least 12 weeks of standardized therapy prior to screening.

2.Refractory Idiopathic inflammatory myopathy (IIM) 2.1.Age 18-70 years. 2.2.Estimated life expectancy ≥ 3 months. 2.3.Documented disease history and diagnosis for ≥ 6 months prior to screening. 2.4.Participants must agree to use effective contraception throughout the study; women of child-bearing potential must have a negative pregnancy test.

2.5.Signed informed consent, agreement to the treatment protocol, and willingness to attend follow-up evaluations per schedule.

2.6.Relevant medical history and clinical manifestations: provide a copy of inpatient records from a tertiary hospital or outpatient records and diagnostic certificates within the last 3 months.

2.7.Fulfillment of the 2017 EULAR/ACR classification criteria for dermatomyositis or polymyositis.

2.8.Inadequate response to, or intolerance of, at least 12 weeks of standardized therapy prior to screening.

3.Refractory Systemic sclerosis (SSc) 3.1.Age 18-70 years. 3.2.Estimated life expectancy ≥ 3 months. 3.3.Documented disease history and diagnosis for ≥ 6 months prior to screening. 3.4.Participants must agree to use effective contraception throughout the study; women of child-bearing potential must have a negative pregnancy test.

3.5.Signed informed consent, agreement to the treatment protocol, and willingness to attend follow-up evaluations per schedule.

3.6.Relevant medical history and clinical manifestations: provide a copy of inpatient records from a tertiary hospital or outpatient records and diagnostic certificates within the last 3 months.

3.7.Fulfillment of the 2013 ACR/EULAR classification criteria for systemic sclerosis, with clinical or radiographic evidence of pulmonary involvement.

3.8.Required laboratory tests, including but not limited to: CBC, urinalysis, ANA, anti-dsDNA, ENA panel, C3/C4, immunoglobulins, etc.

3.9.Classification per current international or domestic standards: the 1980 ACR criteria for SSc OR the 2013 ACR/EULAR criteria for SSc.

3.10.Inadequate response to, or intolerance of, at least 12 weeks of standardized therapy prior to screening.

4.Refractory Pemphigus 4.1.Age 18-70 years. 4.2.Estimated life expectancy ≥ 3 months. 4.3.Documented disease history and diagnosis for ≥ 6 months prior to screening. 4.4.Participants must agree to use effective contraception throughout the study; women of child-bearing potential must have a negative pregnancy test.

4.5.Signed informed consent, agreement to the treatment protocol, and willingness to attend follow-up evaluations per schedule.

4.6.Relevant medical history and clinical manifestations: provide a copy of inpatient records from a tertiary hospital or outpatient records and diagnostic certificates within the last 3 months.

4.7.Fulfillment of at least one clinical manifestation plus one histopathological or immunodiagnostic criterion, OR at least two clinical manifestations plus two immunodiagnostic criteria:

* Clinical manifestations: flaccid cutaneous bullae and fragile blisters that rupture easily, resulting in persistent erosions; mucosal blisters or erosions; positive Nikolsky sign.
* Histopathology: intraepidermal or intraepithelial acantholysis.
* Immunodiagnostic criteria: direct immunofluorescence (DIF) showing intercellular IgG and/or complement deposition in epidermal/epithelial cells of lesional or perilesional normal skin; positive serum anti-epithelial cell antibodies by indirect immunofluorescence; positive serum anti-desmoglein antibodies by ELISA.

4.8.Pemphigus Disease Area Index (PDAI) ≥ 9 (moderate 9-24, severe ≥ 25). 4.9.Inadequate response to, or intolerance of, at least 12 weeks of standardized therapy prior to screening.

5.Refractory Moderate-to-Severe Psoriasis 5.1.Age 18-70 years. 5.2.Estimated life expectancy ≥ 3 months. 5.3.Documented disease history and diagnosis for ≥ 6 months prior to screening. 5.4.Participants must agree to use effective contraception throughout the study; women of child-bearing potential must have a negative pregnancy test.

5.5.Signed informed consent, agreement to the treatment protocol, and willingness to attend follow-up evaluations per schedule.

5.6.Relevant medical history and clinical manifestations: provide a copy of inpatient records from a tertiary hospital or outpatient records and diagnostic certificates within the last 3 months.

5.7.In accordance with the 2023 Chinese Guidelines for the Diagnosis and Treatment of Psoriasis, meets the diagnostic criteria for moderate-to-severe plaque psoriasis: dark-red or infiltrated erythematous plaques covered by white/silvery scales, demonstrating the wax-drip, film, and Auspitz signs.

5.8.At screening: Body Surface Area (BSA) involvement ≥ 10%, Psoriasis Area and Severity Index (PASI) ≥ 10, and static Physician's Global Assessment (sPGA) ≥ 3.

5.9.Inadequate response to, or intolerance of, at least 12 weeks of standardized therapy prior to screening.

6.Refractory Moderate-to-Severe Rheumatoid Arthritis 6.1.Age 18-70 years. 6.2.Estimated life expectancy ≥ 3 months. 6.3.Documented disease history and diagnosis for ≥ 6 months prior to screening. 6.4.Participants must agree to use effective contraception throughout the study; women of child-bearing potential must have a negative pregnancy test.

6.5.Signed informed consent, agreement to the treatment protocol, and willingness to attend follow-up evaluations per schedule.

6.6.Relevant medical history and clinical manifestations: provide a copy of inpatient records from a tertiary hospital or outpatient records and diagnostic certificates within the last 3 months.

6.7.Required laboratory and imaging assessments, including but not limited to: ESR, CRP, rheumatoid factor, ANA, anti-CCP antibodies, and other relevant autoantibodies; bilateral hand/foot radiographs.

6.8.Meets current international or domestic classification criteria: the 1987 ACR criteria for RA OR the 2010 ACR/EULAR criteria for RA.

6.9.Inadequate response to, or intolerance of, at least 12 weeks of standardized therapy prior to screening.

7.Refractory ANCA-Associated Vasculitis/Nephritis 7.1.Age 18-70 years. 7.2.Estimated life expectancy ≥ 3 months. 7.3.Documented disease history and diagnosis for ≥ 6 months prior to screening. 7.4.Participants must agree to use effective contraception throughout the study; women of child-bearing potential must have a negative pregnancy test.

7.5.Signed informed consent, agreement to the treatment protocol, and willingness to attend follow-up evaluations per schedule.

7.6.Relevant medical history and clinical manifestations: provide a copy of inpatient records from a tertiary hospital or outpatient records and diagnostic certificates within the last 3 months.

7.7.Meets the 2022 ACR/EULAR classification criteria for vasculitis. 7.8.Renal biopsy indicating kidney involvement, or clinical manifestations consistent with small-vessel vasculitis together with positive myeloperoxidase (MPO) or proteinase-3 (PR3) antibodies.

7.9.Persistent or newly emerging renal and/or systemic vasculitic manifestations despite maintenance therapy of the same intensity as initial immunosuppressive treatment.

7.10.Inadequate response to, or intolerance of, at least 12 weeks of standardized therapy prior to screening.

Exclusion Criteria:

* (1) Clinically significant (as determined by the investigator) history of cardiac, endocrine, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic, or other major diseases.

  (2) Pregnant or lactating women. (3) History of active tuberculosis (TB) infection within 3 years prior to the screening visit.

  (4) History of traumatic brain injury, altered consciousness, epilepsy, cerebral ischemia, or any cerebrovascular hemorrhagic disorders.

  (5) Prolonged QT interval on ECG or history of severe arrhythmias or other significant cardiac disorders.

  (6) Active infection (excluding uncomplicated urinary tract infection and bacterial pharyngitis).

  (7) Active hepatitis B virus or hepatitis C virus infection. (8) Confirmed positive anti-HIV antibody test. (9) Positive Treponema pallidum antibody test judged by the investigator to be clinically significant.

  (10) Any known or suspected congenital or acquired immunodeficiency that may compromise the subject's immune status.

  (11) Prior treatment with CD19 CAR-T cell therapy or CD19-targeted antibody drugs.

  (12) Prior exposure to any gene therapy. (13) ALT/AST > 3× ULN, or bilirubin > 2.0× ULN, or serum creatinine > 2× ULN, or creatinine clearance < 30 mL/min.

  (14) Any condition that, in the opinion of the investigator, may increase patient risk or interfere with study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-08-18 (Estimated); Study Completion 2027-11-18 (Estimated)

PRIMARY OUTCOMES:
Phase I:Cytokine Release Syndrome (CRS) | 28 days post infusion
  The incidence and severity of Cytokine Release Syndrome (CRS)
Phase I：Immune Effector Cell-Associated Neurotoxicity Syndrome(ICANS) | 28 days post infusion
  The incidence and severity of Immune Effector Cell-Associated Neurotoxicity Syndrome(ICANS)
Phase II: Efficacy:Objective response rate (ORR) | 3 months and 6 months post infusion
  Proportions of subjects achieving Autoimmune Diseases response

SECONDARY OUTCOMES:
AUCS of CAR-T cells [Cell dynamics] | Up to 6 months post infusion
  AUCS is defined as the area under the curve in 6 months
CMAX of CD19 CAR T cells [Cell dynamics] | Up to 6 months post infusion
  CMAX is defined as the highest concentration of CD19 CAR T cells expanded in peripheral blood
TMAX of CD19 CAR T cells [Cell dynamics] | Up to 6 months post infusion
  TMAX is defined as the time to reach the highest concentration
CAR-T proliferation [Cell dynamics] | Up to 6 months post infusion
  the copy number of Senl CAR- T cells in the genomes of PBMC by qPCR method
Pharmacodynamics of CD19 CAR T cells | Up to 6 months post infusion
  IL-6 levels measured by Chemiluminescence method
B cell levels in peripheral blood | Up to 6 months post infusion
  The change of B cell levels in peripheral blood after infusion
SLE:Systemic Lupus Erythematosus Disease Activity Index 2000(SLEDAI-2K) | Up to 6 months post infusion
  The Change of Systemic Lupus Erythematosus Diseases Activity Index, (SLEDAI-2k) from baseline.
  Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) helped standardize outcome measures in SLE and is a clinical tool predominantly used in research to track disease activity and response to therapy.
  SLEDAI score (obtained by adding the individual 24 item scores) ranges from 0 to 105, where the higher the score, the greater the degree of disease activity.
  No Flare (Disease no active): 0-3 Mild or moderate flare ( Mild or moderate Active): 4-12 Severe Flare (Severe Active): ≥ 13
IIM:Remission Rate | Up to 6 months post infusion
  Per the International Myositis Assessment and Clinical Studies Group (IMACS) criteria, complete remission is defined as normalization of all activity measures with no new symptoms, whereas partial remission is defined as improvement of ≥50 % of the baseline abnormal measures.
SSc:modified Rodnan Skin Score (mRSS) | Up to 6 months post infusion
  Skin improvement will be assessed using the modified Rodnan Skin Score (mRSS). A clinically significant improvement is defined as a ≥5-point absolute decrease or a ≥25 % relative reduction from baseline; stability is defined as a change of ≤3 points.
SSc: Pulmonary fibrosis progression | Up to 6 months post infusion
  Pulmonary fibrosis progression is defined as a ≥10 % decline in percent-predicted FVC and/or a ≥15 % decline in percent-predicted DLCO, or evidence of progressive fibrosis on high-resolution chest CT.
Pemphigus:Pemphigus Disease Area Index (PDAI). | Up to 6 months post infusion
  Disease activity will be assessed with the Pemphigus Disease Area Index (PDAI).
  * Complete remission: PDAI = 0 and no new blisters.
  * Partial remission: ≥ 75 % reduction in PDAI from baseline.
  * Treatment failure: < 50 % reduction in PDAI from baseline or appearance of new blisters.
Psoriasis:Psoriasis Area and Severity Index (PASI) | Up to 6 months post infusion
  In accordance with the 2023 Chinese Guidelines for the Diagnosis and Treatment of Psoriasis, treatment response will be evaluated using the Psoriasis Area and Severity Index (PASI)
  * Complete clearance: 100 % improvement in PASI.
  * Almost complete clearance: 90 - 100 % improvement in PASI.
  * Effective response: 75 - 90 % improvement in PASI.
  * Treatment failure: ≤ 50 % improvement in PASI.
RA:IIM:Remission Rate | Up to 6 months post infusion
  Rheumatoid arthritis: Response will be assessed using ACR, EULAR, SDAI, and CDAI criteria, with the goal of achieving disease remission or a response at least equivalent/superior to that afforded by conventional therapy.
ANCA-associated vasculitis/nephritis:Birmingham Vasculitis Activity Score (BVAS) | Up to 6 months post infusion
  ANCA-associated vasculitis/nephritis: According to the 2024 KDIGO Clinical Practice Guideline for the Management of ANCA-Associated Vasculitis, disease outcomes will be evaluated with the Birmingham Vasculitis Activity Score (BVAS). Remission is defined as the absence of active vasculitis and glomerulonephritis (BVAS = 0), and relapse is defined as renewed disease activity after partial or complete remission.

CONTACTS AND LOCATIONS:
Overall Officials: Huirui Wang, M.D., Principal Investigator — Henan Province Engineering Technology Research Center of Immunological Precision Medicine and Artificial Intelligence Application, The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, China
Locations (1):
- Henan Province Engineering Technology Research Center of Immunological Precision Medicine and Artificial Intelligence Application, The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, China, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: No